CLINICAL TRIAL: NCT01768546
Title: Evaluation of Video On-Demand Programming to Prevent Type 2 Diabetes in Adults
Acronym: Project NOT ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UnitedHealth Group (Industry)
Collaborators: Comcast Corporation (Unknown); Dr. Ron Ackermann (Unknown)
Responsible Party: Principal Investigator, Dr. Deneen Vojta, Dr. Deneen Vojta Vice President of Center for Health Reform and Modernization, UnitedHealth Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Project NOT ME 11-351
Record Dates: First submitted 2013-01-09; First posted 2013-01-15 (Estimated); Last update posted 2014-12-19 (Estimated); Status verified 2014-12

CONDITIONS: Pre-diabetes
Keywords: Diabetes Prevention Program; obesity; activity; diabetes
MeSH Terms: conditions — Glucose Intolerance; Obesity; Motor Activity; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Video on Demand (VOD) (Experimental): Virtual Diabetes Prevention Program: All participants will view the 16 Comcast on Demand episodes, weigh themselves, and track their progress weekly. Participants in the VOD arm of the study received access to a paper tracker to track food and activity during the program.
  Interventions: Behavioral: Virtual Diabetes Prevention Program
- Video on Demand Plus (VOD+) (Experimental): Virtual Diabetes Prevention Program: All participants will view the 16 Comcast on Demand episodes, weigh themselves, and track their progress weekly. Participants in the VOD+ arm of the trial received access an interactive tracking and problem solving web portal offered by SparkPeople™ (Cincinnati, Ohio).
  Interventions: Behavioral: Virtual Diabetes Prevention Program; Behavioral: Interactive tracking and problem solving web portal

INTERVENTIONS:
Behavioral: Virtual Diabetes Prevention Program — Participants will view 16 Video On Demand reality based TV episodes that follow 6 adults with pre-diabetes actively participating in a DPP lifestyle intervention.
  Other Names: Lifestyle Change Program
Behavioral: Interactive tracking and problem solving web portal
  Other Names: Web-based lifestyle support
  Arms: Video on Demand Plus (VOD+)

SUMMARY:
Over the past 40 years, diabetes has increased dramatically in parallel with rapid increases in obesity.About 90 to 95% of persons with diabetes have type 2 diabetes, which begins when the body becomes resistant to the hormone insulin. Insulin resistance results from weight gain and physical inactivity, making the vast majority of new cases of type 2 diabetes preventable with lifestyle changes.

After the findings of the Diabetes Prevention Program were released in 2002, the high cost of the lifestyle program prevented it from becoming widely adopted throughout the U.S.

The UnitedHealth Center for Health Reform and Modernization (CHRM) will evaluate the use and effectiveness of a scalable approach for providing lifestyle-based diabetes prevention intervention through Comcast's XFINITY Video-On-Demand (VOD) programming, with additional non-compulsory support from SparkPeopleTM (Cincinnati, Ohio), an interactive tracking and problem solving web portal. By design, this effort will engage adult television viewers and offer them education and resources to support their efforts to achieve levels of weight loss and physical activity which have previously shown to prevent the development of type 2 diabetes. Specifically, we aim to evaluate:

1. Viewing patterns and characteristics of consumers accessing a prevention program via VOD
2. Effectiveness in terms of weight loss achieved
3. Consumers' ratings of overall content

DETAILED DESCRIPTION:
Obesity, pre-diabetes, and diabetes are related diseases that are reaching epidemic proportions in the United States. In order to ultimately control health care costs, employers, private payers and public payers must address this issue with models that effectively identify individuals with these conditions and aggressively intervene to improve compliance with evidence-based care standards.

Project NOT ME leverages a proven model that drives earlier identification, improved individual compliance, better health outcomes, and lower costs for the consumer, the payer and plan sponsors. More specifically, Project NOT ME provides a solution by offering pre-diabetic participants access to a virtual program that includes a reality TV show, an electronic scale and trackers. Project NOT ME is an evidence-based intervention that follows the National Diabetes Prevention Program (DPP). It is designed to enact lifestyle changes that result in a safe reduction in weight, and a reduction in conversion to full blown type-2 diabetes.

Project NOT ME is divided in two parts --

1. Program: For the first 20 weeks, participants work to become more aware of the food they eat, and the amount of exercise they are getting. The Video on Demand episodes educate participants on strategies that are proven to help them make better food choices, and find time in their lives to be more active. During the core program, participants will:

   * Weigh themselves every week using a program-provided electronic scale that automatically records their weight and sends to the study team
   * Log all the food they eat and all the exercise they are getting in a tracker
   * Watch 16 episodes of a captivating reality based TV show that highlights 6 adults participating in the Diabetes Prevention Program.
   * Review weekly online episode summaries.
2. Maintenance Sessions: For the next 32 weeks, participants will practice what they learned in the Core Sessions, continue to track food and exercise, and have access to the television episodes.

ELIGIBILITY:
Inclusion Criteria:

* Told by a doctor, nurse, or other healthcare provider that he/she has prediabetes or is at very high risk for developing type 2 diabetes
* Told by a doctor, nurse or other healthcare provider that he/she has high blood pressure or is receiving prescription medication to treat high blood pressure
* Told by a doctor, nurse or other healthcare provider that he/she has abnormal blood cholesterol or is receiving prescription medication to treat blood cholesterol
* Has a first-degree blood relative (mother, father, brother or sister) who has or had type 2 diabetes
* Is a woman with a personal history of gestational diabetes (diabetes of pregnancy only)

Exclusion Criteria:

* Currently reports a body weight of more than 310 pounds
* Considering bariatric surgery ("stomach stapling" or gastric bypass) in the next 6 months
* Told by a doctor or nurse that they have diabetes (except diabetes of pregnancy alone) or is receiving any form of treatment for diabetes
* Has poorly controlled high blood pressure, typically more than 180/105, that has not been discussed with a healthcare provider
* Is a woman who is currently pregnant or actively planning pregnancy in the next 6 months
* Has chest pain, dizziness, or severe shortness of breath or bodily weakness with even moderate levels of physical exertion such as brisk walking
* Has been told by a doctor or nurse not to increase his/her current level of physical activity or not to attempt weight loss
* Has any other condition, such as advanced heart or lung disease, severe painful arthritis, or another disability that significantly limits physical activities such as brisk walking
* Has any other condition, such as malnutrition or unexplained weight loss in which attempts to lose additional body weight could be unsafe

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 306 (Actual)
Dates: Start 2012-02; Primary Completion 2013-05 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Weight Measure at Week 16 | Baseline - Week 16
  Weight measures will be taken on electronic scales that transmit the weight using GSM/cellular technology at the start of the study, after each weekly episode, at the end of the evaluation period (week 16) and after all maintenance materials have been delivered (month 12). Self-reported weight will also be collected in the pre-study survey, follow-up survey and through SparkPeople.com.

SECONDARY OUTCOMES:
Viewing patterns and characteristics of consumers accessing a prevention program via VOD | Week 16
  The following viewing data will be captured by Comcast and made available to the evaluation team with permission from the study participant: date and title for each episode viewed (date / time stamp for episode initiation, total viewing time, confirmation whether episode was viewed in its entirety or viewed more than once).
Consumers' ratings of overall content | Week 16
  A survey will be be administered at week 16 containing health related and work productivty questions, the perceived usefulness of the content,intent to make changes in behavior and likelihood to recommend the program to others.
Change from Baseline Weight Measure at Month 12 | Baseline and Month 12
  Weight measures will be taken on electronic scales that transmit the weight using GSM/cellular technology at the start of the study, after each weekly episode, at the end of the evaluation period (week 16) and after all maintenance materials have been delivered (month 12). Self-reported weight will also be collected in the pre-study survey, follow-up survey and through SparkPeople.com.

CONTACTS AND LOCATIONS:
Overall Officials: Deneen Vojta, MD, Principal Investigator — UnitedHealth Group